CLINICAL TRIAL: NCT00785902
Title: AtriCure Bipolar Radiofrequency Ablation of Persistent Atrial Fibrillation
Acronym: A
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Other Study IDs: CP2008-1
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AtriCure Bipolar System

SUMMARY:
ABLATE Persistent is a prospective, non-randomized multi-center clinical trial to demonstrate the safety and effectiveness of the AtriCure Bipolar System for treating persistent atrial fibrillation during concomitant on-pump cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age
2. Subject has history of persistent atrial fibrillation as defined by the ACC/AHA/ESC Guidelines
3. Subject is scheduled to undergo elective on-pump cardiac surgical procedure(s) for one or more of the following:

   * Mitral valve repair or replacement
   * Aortic valve repair or replacement
   * Tricuspid valve repair or replacement
   * Coronary Artery Bypass procedures
4. Subject's Left Ventricular Ejection Fraction ≥ 30%
5. Subject is able and willing to provide written informed consent and comply with study requirements
6. Subject has life expectancy of at least 1 year

Exclusion Criteria:

1. Patients with longstanding and continuous AF in which cardioversion has failed or has not been attempted
2. Previous cardiac ablation including catheter ablation, AV-nodal ablation, or surgical Maze procedure
3. Wolff-Parkinson-White syndrome
4. Prior cardiac surgery (Redo)
5. Class IV NYHA heart failure symptoms
6. Prior history of cerebrovascular accidents within 6 months or at any time if there is residual neurological deficit
7. Documented MI within 6 weeks prior to study enrollment
8. Need for emergent cardiac surgery (i.e. cardiogenic shock)
9. Known carotid artery stenosis greater than 80%
10. LA size greater than or equal to 8 cm
11. Current diagnosis of active systemic infection
12. Severe peripheral arterial occlusive disease defined as claudication with minimal exertion
13. Pregnancy or desire to get pregnant within 12-months of the study enrollment
14. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
15. Renal failure requiring dialysis or hepatic failure
16. Requires anti-arrhythmic drug therapy for the treatment of a ventricular arrhythmia
17. Therapy resulting in compromised tissue integrity including: thoracic radiation, chemotherapy, long term treatment with oral or injected steroids, or known connective tissue disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The primary efficacy endpoint for this study is the percent of patients free from AF and off Class I and III antiarrhythmic drugs at 9 months.
The primary safety endpoint is the composite acute major adverse event rate, within 30 days post-procedure or hospital discharge

SECONDARY OUTCOMES:
The secondary efficacy endpoint for this study is the percent of patients free from AF, independent of antiarrhythmic drug status at 9 months
The secondary safety endpoint is the composite 9-month post-procedure major adverse event rate.